CLINICAL TRIAL: NCT03717844
Title: Registry for Adults With Plasma Cell Disorders (PCD's)
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1728
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Amyloidosis; Cryoglobulinemia; Castleman's Disease; Light Chain Deposition Disease; Heavy Chain Deposition Disease; Polyneuropathy Organomegaly Endocrinopathy Monoclonal Gammopathy and Skin Changes; Smoldering Multiple Myeloma; Plasma Cell Leukemia
MeSH Terms: conditions — Multiple Myeloma; Amyloidosis; Cryoglobulinemia; Castleman Disease; POEMS Syndrome; Smoldering Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples will be banked for future research involving adults with PCDs, specifically examining p16INK4a and other markers to be specified in future, separate, IRB-reviewed protocols as specific research questions are identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary purpose of this protocol is to create a registry of patients with plasma cell disorders (PCDs), including for example the cancer multiple myeloma (MM), who complete the assessment, previously known as a "geriatric assessment," as is outlined in this protocol. Secondary objectives include measuring the response rate to participation of patients in this study, assessing patient satisfaction with the questionnaire, and gathering information that would lend support for future research into these types of assessments in patients with PCDs. Additionally the study offers an optional blood draw to look at a genetic marker of aging called p16INK4a (IRB 15-1899, IRB 15-0244).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

1. To create a Registry (to be called the PCD Registry) of PCD patients
2. To have participating patients complete an assessment at enrollment and to repeat the assessment longitudinally over time.

Secondary

1. To gather information, including patterns of patient care, that would lend support for future research in the PCD population. Specific research questions would be explored within separate IRB-reviewed protocols.
2. To bank blood samples for future research involving adults with PCD's, specifically examining p16INK4a and other markers to be specified in future, separate, IRB-approved protocols as specific research questions are identified.

OUTLINE: Patients complete an assessment at baseline and then longitudinally over time which involves a multi-dimensional inter-disciplinary evaluation of a patient's functional status (ability to live independently at home and in the community), co-morbid medical conditions, cognition, psychological status, social functioning and support, medication review, and nutritional status. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients have an outpatient appointment or are hospitalized inpatient at UNC Cancer Hospitals, or affiliated clinic settings or participating sites for the evaluation and management of a PCD.
* Patients have a documented diagnosis of PCD defined as the presence of a monoclonal protein and/or monoclonal plasma cell population. Examples of PCDs include but are not limited to monoclonal gammopathy of uncertain significance; smoldering myeloma; multiple (active) myeloma; plasma cell leukemia; Castleman's disease; amyloidosis; light and/or heavy chain deposition disease; Polyneuropathy, Organomegaly, Endocrinopathy,Monoclonal gammopathy and Skin changes (POEMS) syndrome; and cryoglobulinemia.
* Age ≥18 years.
* Must consent to participation in this study and agree to complete the assessment at baseline and follow-up time points.
* Must be able to read and speak English.

Exclusion Criteria:

* Physical or psychiatric/behavioral illnesses or problems that the treating clinician feels would preclude successful participation in the study.
* There are no imaging or lab studies required to determine eligibility.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients have a documented diagnosis of PCD defined as the presence of a monoclonal protein and/or monoclonal plasma cell population.
  Examples of PCDs include but are not limited to monoclonal gammopathy of uncertain significance; smoldering myeloma; multiple (active) myeloma; plasma cell leukemia; Castleman's disease; amyloidosis; light and/or heavy chain deposition disease; Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal gammopathy and Skin changes (POEMS) syndrome; and cryoglobulinemia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Creation of a Registry of Plasma Cell Disorder (PCD) patients | 10 years
Completion of baseline and longitudinal assessments in PCD patients | 10 years

SECONDARY OUTCOMES:
Creation of information that would lend support for future PCD research | 10 years
  Including patterns of patient care that would lend support for future research in patients with confirmed PCD's.
Response rates of assessment in PCD patients and their satisfaction with the assessment | 10 years
  Done by measuring:
  * percentage of patients contacted who consent to complete the assessment percentage of patients able to complete the self-administered portion of the assessment without assistance
  * the length of time necessary to complete the assessment
  * the variance and number of missing items
  * the percentage of geriatric assessments that contain all three of the following items: Timed Up and Go Assessment, Blessed Orientation-Memor Concentration Test, and the healthcare professional-rated Karnofsky performance status.

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Tuchman, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hospital, Chapel Hill, North Carolina, United States